CLINICAL TRIAL: NCT05111067
Title: Molecular Subtyping of Triple-negative Breast Cancer and African Ancestry-related Immunogenicity
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Obafemi Awolowo University (Other)
Responsible Party: Sponsor
Other Study IDs: 42127
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh frozen Triple-negative breast cancer tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nova scotia TNBC cohort: DNA and whole transcriptome mRNA sequencing, including total mutational burden and microsatellite instability, will be performed using the TruSight Oncology 500 (TSO500) platform (Illumina Canada, Ulc). Transcriptome data will be used to categorize specimens into one of four distinct mRNA subgroups and will be compared between cohorts.
  Interventions: Genetic: DNA and whole transcriptome mRNA sequencing
- Nigerian TNBC cohort: DNA and whole transcriptome mRNA sequencing, including total mutational burden and microsatellite instability, will be performed using the TruSight Oncology 500 (TSO500) platform (Illumina Canada, Ulc). Transcriptome data will be used to categorize specimens into one of four distinct mRNA subgroups and will be compared between cohorts.
  Interventions: Genetic: DNA and whole transcriptome mRNA sequencing

INTERVENTIONS:
Genetic: DNA and whole transcriptome mRNA sequencing — DNA and whole transcriptome mRNA sequencing, including total mutational burden and microsatellite instability, will be performed using the TruSight Oncology 500 (TSO500) platform (Illumina Canada, Ulc).

SUMMARY:
Triple-negative breast cancer (TNBC) is a heterogeneous disease that is associated with a younger age of onset, worse stage matched-outcomes, and women of African ancestry in North America. A higher incidence of TNBC is also seen in West Africa, despite unique environmental, socioeconomic and modifiable risk factors. Transcriptome analysis of TNBC has delineated four distinct subgroups with therapeutic and prognostic significance. With further characterization, important regional differences have emerged between populations of African vs. European ancestry. These differences may have significant implications for the efficacy of novel TNBC-targeted therapy and need to be further evaluated. Transcriptional data on TNBC in sub-Saharan African also offers the opportunity to evaluate the relationship between breast cancer phenotype and ancestry-linked differences in the tumor-immune microenvironment.

DETAILED DESCRIPTION:
This study seeks to characterize the mRNA profile of TNBC in Nigeria and compare to a reference population in Nova Scotia. Insight into the unique tumor-immune profile of TNBC in Nigeria and the link between the West African-linked Duffy-antigen receptor for chemokines (DARC) and TNBC subtype will be explored for the first time.

Fresh frozen TNBC tissue from the African Research Group for Oncology (ARGO) and Dalhousie/NSHA breast cancer biobanks' will be processing and analyzed by the Genomics Core Facility at Dalhousie University. Clinical data is prospectively collected with specimen acquisition in the ARGO biobank. For the Dalhousie /NSHA biobank, clinical data will be retrospectively gathered from the medical record and migrated to an electronic database for prospective collection during the course of the study. Both cohorts of specimens will be run through DNA and whole transcriptome (mRNA) sequencing on the TSO500 platform (Illumina Ulc.). The tumor-immune microenvironment will be compared between cohorts and by mRNA cluster using the transcriptional signatures for 22 leukocyte populations and immune-regulating proteins CTLA-4 and PD-L1. Finally, tumor expression of DARC will be generated from the transcriptome data that will allow for an assessment of the relationship between DARC expression, TNBC mRNA clusters, and sociodemographic variables (i.e. race/ancestry, gender). Whole transcriptome data from The Cancer Genome Atlas will be pulled as the third cohort, including 55 TNBC specimens from African Americans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Triple-negative breast cancer

Exclusion Criteria:

* No diagnosis of Triple-negative breast cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Biological samples acquired from patient's with Triple-negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
DNA and mRNA sequencing | 3 years
Duffy-antigen receptor for chemokines | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No